CLINICAL TRIAL: NCT04156165
Title: BEEF The Effect of High vs. Moderate Protein Consumption on Human Health - With Beef as Major Source of Protein
Brief Title: The Effect of High vs. Moderate Protein Consumption on Human Health
Acronym: BEEF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Copenhagen (Other)
Collaborators: US National Cattlemen´s Association (Unknown); Danish Agriculture and Food Counsel (Unknown)
Responsible Party: Principal Investigator, Arne Astrup, Professor. Dr.Med, University of Copenhagen
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Treatment
Other Study IDs: B-352; H-19041921 (Registry Identifier: Danish Ethical Committee)
Record Dates: First submitted 2019-11-01; First posted 2019-11-07 (Actual); Last update posted 2021-11-01 (Actual); Status verified 2021-10

CONDITIONS: Weight Loss; Metabolism and Nutrition Disorder; Obesity
Keywords: Body composition; Metabolism
MeSH Terms: conditions — Weight Loss; Nutrition Disorders; Obesity | interventions — Diet, High-Protein

STUDY DESIGN:
Intervention Model Description: 2x2 factorial intervention trial with two and two arms
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- VLCD-Control (Active Comparator): Very low calorie diet, 600 kcal pr day for eight weeks.
  Interventions: Dietary Supplement: VLCD-Control
- VLCD-Active (Experimental): Very low calorie diet plus additional 25 g protein powder, 700 kcal pr day for eight weeks.
  Interventions: Dietary Supplement: VLCD-Active
- Maintenance-Control (Active Comparator): 12-week weight maintenance diets: Moderate protein weight maintenance diet (MP-WMD): Recommended healthy diet including 25 g beef daily.
  The diet is ad libitum and will be high in fibre (40 g/10 MJ) and whole grain (150 g/day) and allow inclusion of free/added sugar up to the recommended level (<10E% sugar).
  Interventions: Other: Maintenance-Control
- Maintenance-Active (Experimental): 12-week weight maintenance diets: High protein weight maintenance diet (HP-WMD): The macronutrient distribution will be 25 energy percentage (E%) from protein, 45 E% from carbohydrate and 30 E% from fat. The diet will include 150 g beef as a daily source of protein, The diet is ad libitum and will be high in fibre (40 g/10 MJ) and whole grain (150 g/day) and allow inclusion of free/added sugar up to the recommended level (<10E% sugar).
  Interventions: Other: Maintenance-Active

INTERVENTIONS:
Dietary Supplement: VLCD-Active — Lighter life formula products supplied to subjects, four sachets pr day. Dietetic advise given regularly.
  Other Names: High protein VLCD
  Arms: VLCD-Active
Other: Maintenance-Active — Weight loss maintenance diet with high protein and low glycemic index and load, high in fiber and whole grain, daily including 150 g minced beef.
  Other Names: High protein diet
  Arms: Maintenance-Active
Dietary Supplement: VLCD-Control — Lighter life VLCD products
  Other Names: Moderat protein VLCD
  Arms: VLCD-Control
Other: Maintenance-Control — Weight loss maintenance diet with moderate protein and low glycemic index and load, high in fiber and whole grain, daily including 25 g minced beef.
  Other Names: Moderate protein diet
  Arms: Maintenance-Control

SUMMARY:
The study will be conducted as a parallel randomized controlled intervention trial, initiated by eight weeks rapid weight loss with one of two VLCDs, one week of reintroducing regular foods, and 12 weeks with one of two different ad libitum diets; in total 21 weeks. The study will be blinded for the statistician. Due to obvious different dietary intakes in the two diets, subjects cannot be blinded and neither the study personnel. As the study includes different dietary recommendations the registered clinical dietician advising the subjects cannot be blinded either.

In total 110 overweight and obese volunteers will be included.

ELIGIBILITY:
Inclusion Criteria:

* Healthy men or women
* Age, 18-65 years
* Overweight or grade I-II obesity (BMI 28-40.0 kg/m2)
* Provided voluntary written informed consent

Exclusion Criteria (main:

* Weight changes ± 5% in the last three months
* Vegetarian, vegan
* Pregnancy or lactation, pregnancy within the past 12 month or plans to become pregnant during the study
* History or diagnosis of diabetes
* History or diagnosis of heart, liver or kidney disease
* History or diagnosis of eating disorders
* Chronic diseases e.g. cancer within the past 5 years (except adequately-treated localized basal cell skin cancer)
* Simultaneous blood donation for other purpose than this study
* Simultaneous participation in other clinical intervention studies
* Use of drugs, that in the opinion of the medically responsible investigator, are likely to affect the outcomes of the study
* Any other condition that judged by the investigator may interfere with the adherence to the study protocol

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 110 (Actual)
Dates: Start 2019-11-01 (Actual); Primary Completion 2020-11-10 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
Body weight | up to week 21
  The subjects will be instructed to stand in the middle of the platform of the scale with a straight neck and eyes looking straight ahead, whilst distributing their weight evenly on both feet. Two measurements are made when the scale has stabilized and both results are noted to the nearest 0.1 kg. The average of the two measurements is used in further analysis.

SECONDARY OUTCOMES:
Body composition | up to week 21
  Body composition will be assessed by DXA as whole body scan
Glucose metabolism | up to week 21
  Measurements of fasting glucose, insulin, HbA1c
Inflammation | Up to week 21
  Measurements of fasting CRP, plasma lipids
Fecal samples | Up to week 21
  Measurement of microbiota (bacteria strains present in feces) and metabolomics markers
Resting metabolic rate | Up to week 21
  Resting metabolic rate will be measured by indirect calorimetry, using a ventilated hood system as described by the manufacture
Endocrine disruptors | Up to week 21
  Measurement of fasting T3 and T4
Height | Week 0
  The participant will be instructed to remove shoes and asked to stand erect with their back to the wall-mounted stadiometer, with the back of their head, back, and buttocks touching the stadiometer. The participant will be further instructed to look straight ahead and keep arms relaxed and hanging loosely alongside their body and to inhale deeply. The reading on the stadiometer will be performed before the participant exhales. Two measurements are made and both results are recorded in centimeters to the nearest 0.5 of a centimeter. The average of the two measurements is used in further analysis.
Waist circumference | Up to week 21
  The measurement of waist circumference will be performed in a fasting condition with an empty bladder. The measure is done with a with a no-elastic tape measure mid-way between the lower rib and iliac crest (top of the hip bone) at the end of expiration with the participant in a standing position with their weight distributed evenly on both feet. Two measurements are made and both results are noted to the nearest 0.5 cm and the average of the two measurements is used in further analysis.
Hip circumference | Up to week 21
  The measurement of hip circumference will be measured in a fasting condition with an empty bladder. The measure is done with a tape measure at the widest point between the hips and buttocks observed from the front at the end of expiration with the participant in a standing position with their weight distributed evenly on both feet. Two measurements are made and both results are noted to the nearest 0.5 cm and the average of the two measurements is used in further analysis.
Blood pressure | Up to week 21
  Systolic and diastolic blood pressure will be measured using a validated automatic device with an appropriate arm cuff after 5-10 min rest in a resting position

OTHER OUTCOMES:
Initial glucose metabolism | Up to week 21
  To investigate the effect of initial glucose metabolism on the response to high vs. moderate protein diet on weight maintenance.
Initial microbiota | Up to week 21
  Statistical investigation of the effect of initial microbiota assessed by fecal sample on weight change
Initial body composition | Up to week 21
  Statistical investigation of the effect of initial body composition assessed by DXA scan on weight change.
Physical activity and sleep | Up to week 21
  Physical activity and sleep patterns will be measured by an accelerometer (ActiGraph GT3X+) in the 7 days/8 nights
Perceived stress | Up to week 21
  Assessed by Perceived Stress Scale questionnaire
Life quality | Up to week 21
  Assessed by SF-36 questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Arne Astrup, Professor, Principal Investigator — Department of Nutrition, Exercise and Sports, UCPH
Locations (1):
- University of Copenhagen, Frederiksberg, DK, Denmark

REFERENCES:
- [Derived] Magkos F, Hjorth MF, Asping S, Rosenkrans MI, Rasmussen SI, Ritz C, Sjodin A, Geiker NRW. A protein-supplemented very-low-calorie diet does not mitigate reductions in lean mass and resting metabolic rate in subjects with overweight or obesity: A randomized controlled trial. Clin Nutr. 2021 Dec;40(12):5726-5733. doi: 10.1016/j.clnu.2021.10.006. Epub 2021 Oct 18. PMID 34749132